CLINICAL TRIAL: NCT04567537
Title: Ablative Fractional Laser Treatment for the Improvement of Hypertrophic Scars and Scleroderma: a Prospective Cohort Study
Brief Title: Laser Treatment for the Improvement of Scars and Scleroderma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment has been slow and we are prioritizing other studies.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Dieter Manstein, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019P002156
Record Dates: First submitted 2020-09-11; First posted 2020-09-28 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Scars; Scleroderma
Keywords: Scar; Scleroderma; Laser
MeSH Terms: conditions — Cicatrix; Scleroderma, Diffuse | interventions — Laser Therapy

STUDY DESIGN:
Intervention Model Description: The investigators will be performing a prospective cohort study, where the entire lesion will receive laser treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Scars (Active Comparator): The entire hypertrophic scar will receive laser treatment only.
  Interventions: Device: Laser Treatment
- Scleroderma (Active Comparator): The entire lesion will receive laser treatment.
  Interventions: Device: Laser Treatment

INTERVENTIONS:
Device: Laser Treatment — Patients will receive three laser treatments at one-month intervals.

SUMMARY:
In this study, the investigators seek to evaluate the effects of a laser treatment on the redistribution/regeneration of collagen on the clinical, microscopic, and molecular profiles of hypertrophic scars and scleroderma.

DETAILED DESCRIPTION:
This study is designed to evaluate the efficacy of laser treatment for the improvement of the clinical appearance of disorders of collagen metabolism, including hypertrophic scars and scleroderma. The investigators will be performing a prospective cohort study. The entire lesion will receive laser treatment only.

The investigators plan to have 20 patients (10 patients with hypertrophic scars and 10 patients with scleroderma) complete the study.

Subjects must be equal to greater than 18 years old, but may be any gender or Fitzpatrick skin type. They must have one of the following: at least one extragenital hypertrophic scar, or at least one extragenital area of scleroderma . Subjects must not have received any prescription or in-clinic medications or treatments, such as intralesional corticosteroids or excision, on the eligible scars/scleroderma in the previous 3 months. Those on anti-inflammatory or immunosuppressive medications will also be excluded.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be able and willing to provide written informed consent and comply with the requirements of the study protocol;
2. In good general health, based on answers provided during the screening visit;
3. Subject must be able to read and understand English;
4. Any gender and any Fitzpatrick skin type;
5. Age equal to or greater than 18 years old;
6. Subjects in the hypertrophic scar branch must have at least one extragenital hypertrophic scar (defined as abnormal proliferation of scar tissue that forms at the site of cutaneous injury and does not regress and grows beyond the original margins of the scar) large enough to treat for both the control and experimental arm (at least 4cm in length for spit scar treatment) or two similar hypertrophic scars (at least 4cm2 for each);
7. Subjects in the scleroderma branch must have eligible extragenital lesions; large enough to treat for both the control and experimental arm or two similar scleroderma areas (at least 4cm2 area for each);

Exclusion Criteria:

1. Participation in another investigational drug or device clinical trial in the past 30 days;
2. Are pregnant or lactating;
3. Use of any prescription or in-clinic medications or treatments, such as intralesional corticosteroids or excision, on the eligible scars/scleroderma in the previous 3 months;
4. History of allergic reaction to topical or local anesthesia;
5. Regular intake of high doses of anti-inflammatory drugs (aspirin >81 mg/day, ibuprofen, corticosteroids, etc.) or immunosuppressive drugs;
6. Clinically significant abnormal findings or conditions which might, in the opinion of the Investigator, interfere with study evaluations or pose a risk to subject safety during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Physician's Global Assessment Scale | baseline, pre-intervention
  A score of 0 denotes "No evidence of disease, 100% improvement" and "Completely clear." A score of 1 denotes "Very significant clearance (≥90% to 100%); only traces of disease remain" and "Almost Clear." A score of 2 denotes "Significant improvement(≥75% to < 90%); some evidence of disease remains" and "Marked Improvement." A score of 3 denotes "Intermediate between slight and marked improvement (≥50% to <75%)" and "Moderate Improvement." A score of 4 denotes "Some improvement (≥25% to <50%); significant evidence of disease remains" and "Slight Improvement ." A score of 5 denotes "Disease has not changed from baseline (+ or - <25%)" and "No Change." A score of 6 denotes "Disease is worse than at baseline by ≥25% or more" and "Worse."
Physician's Global Assessment Scale | 1 month after baseline
  A score of 0 denotes "No evidence of disease, 100% improvement" and "Completely clear." A score of 1 denotes "Very significant clearance (≥90% to 100%); only traces of disease remain" and "Almost Clear." A score of 2 denotes "Significant improvement(≥75% to < 90%); some evidence of disease remains" and "Marked Improvement." A score of 3 denotes "Intermediate between slight and marked improvement (≥50% to <75%)" and "Moderate Improvement." A score of 4 denotes "Some improvement (≥25% to <50%); significant evidence of disease remains" and "Slight Improvement ." A score of 5 denotes "Disease has not changed from baseline (+ or - <25%)" and "No Change." A score of 6 denotes "Disease is worse than at baseline by ≥25% or more" and "Worse."
Physician's Global Assessment Scale | 2 months after baseline
  A score of 0 denotes "No evidence of disease, 100% improvement" and "Completely clear." A score of 1 denotes "Very significant clearance (≥90% to 100%); only traces of disease remain" and "Almost Clear." A score of 2 denotes "Significant improvement(≥75% to < 90%); some evidence of disease remains" and "Marked Improvement." A score of 3 denotes "Intermediate between slight and marked improvement (≥50% to <75%)" and "Moderate Improvement." A score of 4 denotes "Some improvement (≥25% to <50%); significant evidence of disease remains" and "Slight Improvement ." A score of 5 denotes "Disease has not changed from baseline (+ or - <25%)" and "No Change." A score of 6 denotes "Disease is worse than at baseline by ≥25% or more" and "Worse."
Physician's Global Assessment Scale | 3 months after baseline
  A score of 0 denotes "No evidence of disease, 100% improvement" and "Completely clear." A score of 1 denotes "Very significant clearance (≥90% to 100%); only traces of disease remain" and "Almost Clear." A score of 2 denotes "Significant improvement(≥75% to < 90%); some evidence of disease remains" and "Marked Improvement." A score of 3 denotes "Intermediate between slight and marked improvement (≥50% to <75%)" and "Moderate Improvement." A score of 4 denotes "Some improvement (≥25% to <50%); significant evidence of disease remains" and "Slight Improvement ." A score of 5 denotes "Disease has not changed from baseline (+ or - <25%)" and "No Change." A score of 6 denotes "Disease is worse than at baseline by ≥25% or more" and "Worse."
Physician's Global Assessment Scale | 4 months after baseline
  A score of 0 denotes "No evidence of disease, 100% improvement" and "Completely clear." A score of 1 denotes "Very significant clearance (≥90% to 100%); only traces of disease remain" and "Almost Clear." A score of 2 denotes "Significant improvement(≥75% to < 90%); some evidence of disease remains" and "Marked Improvement." A score of 3 denotes "Intermediate between slight and marked improvement (≥50% to <75%)" and "Moderate Improvement." A score of 4 denotes "Some improvement (≥25% to <50%); significant evidence of disease remains" and "Slight Improvement ." A score of 5 denotes "Disease has not changed from baseline (+ or - <25%)" and "No Change." A score of 6 denotes "Disease is worse than at baseline by ≥25% or more" and "Worse."
Physician's Global Assessment Scale | Up to 1 year after baseline
  A score of 0 denotes "No evidence of disease, 100% improvement" and "Completely clear." A score of 1 denotes "Very significant clearance (≥90% to 100%); only traces of disease remain" and "Almost Clear." A score of 2 denotes "Significant improvement(≥75% to < 90%); some evidence of disease remains" and "Marked Improvement." A score of 3 denotes "Intermediate between slight and marked improvement (≥50% to <75%)" and "Moderate Improvement." A score of 4 denotes "Some improvement (≥25% to <50%); significant evidence of disease remains" and "Slight Improvement ." A score of 5 denotes "Disease has not changed from baseline (+ or - <25%)" and "No Change." A score of 6 denotes "Disease is worse than at baseline by ≥25% or more" and "Worse."

SECONDARY OUTCOMES:
Mouth Handicap in Systemic Sclerosis scale | Compare baseline to post-procedural
  To assess facial scleroderma
Vancouver Scar Scale | Compare baseline to post-procedural
  To assess all scars, facial and non-facial
Range of Motion Evaluation | Compare baseline to post-procedural
  For non-facial scleroderma to evaluate range of motion of the joint by assessing flexion, extension, supination, and pronation using a goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Manstein, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Clinical Unit for Research Trials & Outcomes in Skin, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.